CLINICAL TRIAL: NCT06728657
Title: A Phase II Randomized Trial of Preoperative Hypofractionated Radiotherapy (HFRT) Compared to Personalized Hyperfractionated Stereotactic Adaptive Radiotherapy (PULSAR), Combined With Chemotherapy and PD-1 Monoclonal Antibody for Locally Advanced Gastroesophageal Junction/Proximal Gastric Adenocarcinoma
Brief Title: Preoperative HFRT Verses PULSAR for Locally Advanced GEJ or Proximal Gastric Adenocarcinoma
Acronym: TORCH-G
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficult in recruiting participants
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Professor, Chief Physician, Head of Department of Radiation Oncology, Fudan University Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-2024-251-3805
Record Dates: First submitted 2024-12-01; First posted 2024-12-11 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Stomach Adenocarcinoma; Gastro-esophageal Junction Cancer
Keywords: radiotherapy; PD-1 inhibitors; chemotherapy; locally advanced; gastrectomy; neoadjuvant; hypofractionated radiotherapy
MeSH Terms: interventions — spartalizumab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- HFRT (Experimental): Participants will receive upfront hypofractionated radiotherapy (HFRT) of the primary lesion and positive lymph nodes (24 Gy/6 fractions). Afterwards, systemic therapy consisted of CAPOX and PD-1 antibodies will be administered every three weeks, for at least 3 cycles. Then, reassessment will be performed within 4 weeks afterwards. For resectable participants, surgical resections of primary lesion will be performed. Postoperative treatment will be determined by the investigators. For unresectable or inoperable participants, the subsequent treatment will be determined by investigators or MDT.
  Interventions: Radiation: HFRT targeted to the primary lesion and positive lymph nodes; Drug: Anti-PD-1 monoclonal antibody; Drug: Chemotherapy; Procedure: R0 total/subtotal gastrectomy with D2 lymphadenectomy
- PULSAR (Experimental): Participants will receive treatment every three weeks, for at least 3 cycles. Each cycle of treatment consists of irradiation (6 Gy/1 fraction) to the primary lesion and positive lymph nodes on day 1, and systemic therapy consisted of CAPOX and PD-1 antibodies will be administered on day 2. Then, reassessment was performed within 4 weeks afterwards. For resectable participants, surgical resections of primary lesion will be performed. Postoperative treatment will be determined by the investigators. For unresectable or inoperable participants, the subsequent treatment will be determined by investigators or MDT.
  Interventions: Radiation: PULSAR targeted to the primary lesion and positive lymph nodes; Drug: Anti-PD-1 monoclonal antibody; Drug: Chemotherapy; Procedure: R0 total/subtotal gastrectomy with D2 lymphadenectomy

INTERVENTIONS:
Radiation: HFRT targeted to the primary lesion and positive lymph nodes — Hypofractionated radiotherapy (HFRT) targeted to the primary lesion and positive lymph nodes (4Gy × 6 fractions)
  Arms: HFRT
Radiation: PULSAR targeted to the primary lesion and positive lymph nodes — Irradiation targeted to the primary lesion and positive lymph nodes (6 Gy/1 fraction)
  Arms: PULSAR
Drug: Anti-PD-1 monoclonal antibody — The anti-PD-1 mAb is used on day 1 along with each cycle of chemotherapy. There are no restrictions on the choice of anti-PD-1 mAb. Patients can choose commonly used accessible monoclonal antibodies based on their personal preferences and financial status. The commonly used anti-PD-1 mAb usages are as follows: Nivolumab, 360mg solution intravenously once daily, Q3W; OR Pembrolizumab/Sintilimab, 200mg solution intravenously once daily, Q3W.
Drug: Chemotherapy — CAPOX: Capecitabine 1000 mg/m2 twice a day, days 1-14 and oxaliplatin 130 mg/m2, day 1, every 3 weeks
Procedure: R0 total/subtotal gastrectomy with D2 lymphadenectomy — For resectable participants, gastrectomy with standard D2 lymphadenectomy is commonly used. The type of gastrectomy performed depends on the location and extent of the primary lesion.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of the multimodal treatment, which includes radiotherapy, chemotherapy and anti-PD-1 immunotherapy. The trial is designed using a pick-the-winner strategy.

The main questions it aims to answer are:

1. If the multimodal treatment will improve the pCR rate.
2. If the multimodal treatment can be performed safely.
3. Hypofractionated radiotherapy (HFRT) or personalized hyperfractionated stereotactic adaptive radiotherapy (PULSAR), which pattern of radiotherapy can better synergize with immunotherapy.

Participants will receive HFRT or PULSAR for the primary lesion and positive lymph nodes, combined with CAPOX and anti-PD-1 immunotherapy. Then, reassessment will be performed within 4 weeks afterwards. For resectable participants, surgical resections will be performed. Postoperative treatment will be determined by the investigators. For unresectable or inoperable participants, the subsequent treatment will be determined by investigators or MDT.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed adenocarcinoma of proximal stomach (G) or gastroesophageal junction (GEJ) (excluding Siewert type I).
* Potentially resectable, cT3-4aN+M0 or cT4bNanyM0.
* Exclusion of peritoneal metastasis through laparoscopic exploration or FAPI PET/CT.
* The status of HER2, MMR, EBER is clear.
* Male or female. Patient age ≥ 18 years and ≤ 75 years.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 or 1.
* Physical state or organ function can tolerate the planned treatment of the study protocol.
* No previous surgery or antitumor therapies, including chemotherapy, radiotherapy, or immunotherapy, were administered.
* Patients agree to sign written informed consent before recruitment.

Exclusion Criteria:

* Pregnancy or breastfeeding women.
* History of other malignancies within 5 years.
* Serious medical illness, such as severe mental disorders, cardiac disease, uncontrolled infection, etc.
* Immunodeficiency disease or long-term using of immunosuppressive agents.
* Allergic to any component of the therapy.
* Any other condition or disease that is not suitable to take the therapy included in the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete regression (pCR) rate | 6 months after the enrollment of the last subject
  Proportion of patients who attain pCR after preoperative treatment.

SECONDARY OUTCOMES:
R0 resection rate | 6 months after the enrollment of the last subject
  Proportion of patients who achieve R0 resection.
Objective response rate (ORR) | 6 months after the recruitment of the last subject
  Proportion of patients with complete response (CR) or partial response (PR) to preoperative therapy. ORR will be evaluated using RESIST1.1
Event-free survival (EFS) | 36 months after the enrollment of the last subject
  EFS is defined as the time interval from enrollment to an event which includes disease progression, discontinuation of the treatment for any reason, or death.
Overall survival (OS) | 36 months after the enrollment of the last subject
  OS is defined as the time interval from enrollment to death of any reason or censoring.
Toxicities | From the time of enrollment, assessed up to 28 days after the last dose of study therapy
  Number of participants with treatment-related adverse events (TrAEs) reported between the first dose and 28 days after the last dose of study therapy as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 5.0.
Surgical morbidity | During or one month after surgery
  Surgery related adverse events (SRAEs) refer to complications which happen during or one month after surgery. Severe complications after surgery will be documented and classified by Clavien-Dindo classification, such as abdominal or GI tract bleeding, anastomotic fistula, pancreatic fistula of grade B or above, and incision complications (infection, bleeding, rupture).
Surgical mortality | During or one month after surgery
  Death from any cause within 30 days of the date of surgery will be considered a surgical mortality death.

OTHER OUTCOMES:
To measure changes in tumor immune microenvironment (TIME) by single-cell sequencing before and after protocol therapy and correlate with the efficacy of the protocol therapy | 36 months after the recruitment of the last subject
The association of baseline PD-L1 CPS, TMB, MSI/MMR status, and EBER status with the efficacy of the protocol therapy | 36 months after the enrollment of the last subject
To study the association between gut microbiota and the efficacy of the protocol therapy | 36 months after the enrollment of the last subject

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No